CLINICAL TRIAL: NCT03473171
Title: Implementation of Nasal Non-Invasive Ventilation With a RAM Cannula in the Inpatient /Outpatient Setting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, James M. Stark, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-17-0708
Record Dates: First submitted 2018-03-14; First posted 2018-03-22 (Actual); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Chronic Respiratory Failure
Keywords: nasal non-invasive ventilation; RAM Cannula; Pediatric Complex Care; Tracheostomy Avoidance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Nasal non-invasive ventilation with RAM cannula (Experimental)
  Interventions: Device: Nasal non-invasive ventilation with RAM cannula

INTERVENTIONS:
Device: Nasal non-invasive ventilation with RAM cannula — Pediatric Pulmonary Team will be consulted on inpatient or outpatient patients that fail to wean from chronic respiratory support (CPAP, BiPAP, High flow Nasal Cannula) in whom long-term ventilation is considered. Pediatric Pulmonary Team, as a consultant, will consider patient history, physical examination, previous imaging and laboratories and previous attempts to wean from respiratory support and causes of failure to wean. The Pulmonary team will determine which patients would potentially benefit from use of NIV/RAM-NC for long-term respiratory support and will recommend initiation of NIV/RAM-NC.

SUMMARY:
The purpose of this study is to implement a standardized protocol to initiate nasal non-invasive ventilation with RAM nasal cannula (NIV/RAM-NC) with Trilogy mechanical ventilator at Children Memorial Hospital inpatient and outpatient sites, as well as to explore the side effects and complications associated with the use of NIV/RAM-NC in children.

ELIGIBILITY:
Inclusion Criteria:

* Children admitted to the Children Memorial Hermann Hospital and consulted to Pediatric Pulmonary Service for initiation of NIV/RAM-NC both at the inpatient and outpatient sites.
* Children who fail to wean from chronic respiratory support (CPAP, BiPAP, HFNC) in whom long-term ventilation is considered between 10/2016 - 10/2017 will be included.

Exclusion Criteria:

* Children with minimal setting (CPAP < 5cmH2O, HFNC < 3LPM) able to be weaned to regular nasal cannula.
* Patients with upper airway obstruction that may be candidates for surgical procedure will be excluded.

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfredo De Jesus Rojas, MD, FAAP, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nasal Non-invasive Ventilation With RAM Cannula
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nasal Non-invasive Ventilation With RAM Cannula
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.92 (7.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 3
  Caucasian | 1
  Hispanic | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Assessed by Number of Participants Who Had Complications
Description: Complications include respiratory failure, tachypnea, hypercapnia, hypoxemia, air trapping or hyperexpansion.
Time Frame: 7 days after starting the RAM cannula
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Non-invasive Ventilation With RAM Cannula
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Nasal Non-invasive Ventilation With RAM Cannula
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT03473171/Prot_SAP_000.pdf